CLINICAL TRIAL: NCT05278026
Title: Cohort Study of Heart Failure With Preserved Ejection Fraction in Chinese Han
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ChiHFpEF-Cohort
Record Dates: First submitted 2021-11-17; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
Keywords: Cardiovascular diseases; Diastolic dysfunction;Systolic dysfunction; Heart failure; Risk factor
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFrEF: heart failure with reduced ejection fraction
  Interventions: Other: guideline recommended routine treatment
- HFpEF: heart failure with preserved ejection fraction
  Interventions: Other: guideline recommended routine treatment
- nonfailing control: patients without heart failure
  Interventions: Other: guideline recommended routine treatment

INTERVENTIONS:
Other: guideline recommended routine treatment

SUMMARY:
To analyze factors contributing to the development and prognosis of heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
Based on previous studies on development of heart failure with preserved ejection fraction (HFpEF), racial/ethnical background should be underscored when evaluating risk f actors for HFpEF incidence. As the ageing population increases sharply in China, HFpEF represents the dominant phenotype of all patients diagnosed with heart failure. In this cohort study, the investigators evaluated exposures or risk factors for HFpEF in Chinese Han patients with cardiovascular diseases (CVD). Our study may provide preventive and therapeutic targets for HFpEF in Chinese CVD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CVD, defined as at least one diagnosis of coronary heart disease, hypertension, type 2 diabetes or cardiomyopathy. The definition of coronary heart disease was stenosis of the main coronary arteries ≥ 50% using percutaneous coronary angiography or coronary computed tomography angiography findings. The definition of hypertension was systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg or pharmacological treatment. The definition of type 2 diabetes was fasting blood glucose ≥ 7.0 mmol/L, random blood glucose ≥ 11.1 mmol/L and HbA1c > 6.5% or the or the use of hypoglycaemic medications. Cardiomyopathy was defined as the presence of cardiac insufficiency in patients with dilated cardiomyopathy suggested by percutaneous coronary angiography or coronary CT angiography use of hypoglycaemic medications.

Exclusion Criteria:

* primary diagnoses of atherosclerosis (stenosis of the main coronary arteries < 50%), congenital heart diseases, arrhythmia, lung diseases, aortic dissection, peripheral vascular diseases, pericardial diseases, myocarditis, hypertrophic cardiomyopathy, heart valvular diseases, cardiophobia, costal chondritis, shock, thyroid diseases, infection or concomitant liver or renal dysfunction.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects were enrolled from Nanjing First Hospital, a public tertiary care university hospital in Nanjing, China.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
One minute sit-to-stand test (1-min STST) | up to 4 weeks
  Briefly, each subject was instructed in sitting position to extend both knees at the same time, starting from a 90° knee flexion position to a 180° extension, which works the thigh muscles, and especially the quadriceps.
Worsening of heart failure (HF) | an average of 1 year
  worsening of symptoms defined as either failure to improve (persistent symptoms and signs of acute HF during treatment) or recurrent symptoms and signs of acute HF, pulmonary edema, or cardiogenic shock after initial stabilization , either of which requiring increased use of diuretics (as outpatient or inpatient), addition of a new intravenous therapy (diuretics, inotrope, or vasodilator) or mechanical support
Hospitalization due to worsening of heart failure (HF) | an average of 1 year
  hospitalization due to worsening HF requiring intravenous pharmacological agents (inotrope or vasodilator), mechanical ventilation, mechanical support or ultra- filtration, hemofiltration, or dialysis

SECONDARY OUTCOMES:
all-cause and cardiogenic deaths | an average of 1 year
  all-cause and cardiogenic deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lp(a) [Lipoprotein(a)]-Related Risk of Heart Failure Is Evident in Whites but Not in Other Racial/Ethnic Groups — https://pubmed.ncbi.nlm.nih.gov/30354212/
- See also: Race/Ethnic Differences in Outcomes Among Hospitalized Medicare Patients With Heart Failure and Preserved Ejection Fraction — https://pubmed.ncbi.nlm.nih.gov/28501527/
- See also: Racial Differences in Characteristics and Outcomes of Patients With Heart Failure and Preserved Ejection Fraction in the Treatment of Preserved Cardiac Function Heart Failure Trial — https://pubmed.ncbi.nlm.nih.gov/29664406/